CLINICAL TRIAL: NCT05843162
Title: A Multi-center, Randomized, Open-label, Active Comparator-controlled, Phase 4 Clinical Trial to Evaluate the Blood Pressure Control of Telmisartan or Losartan in Essential Hypertensive Patients With Metabolic Syndrome
Brief Title: A Clinical Trial to Evaluate the Blood Pressure Control of Telmisartan or Losartan in Essential Hypertensive Patients With Metabolic Syndrome
Acronym: PRISTINE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B115_01HT/MS2201
Record Dates: First submitted 2023-03-09; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Essential Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Essential Hypertension; Metabolic Syndrome | interventions — Telmisartan; Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan (Experimental): Telmitrend Tab.(Telmisartan) 40mg(80mg) + Anydipine-S(S-amlodipine) Tab. 2.5mg
  Interventions: Drug: Telmisartan
- Losartan (Active Comparator): Cozaar Tab.(Losartan) 50mg(100mg) + Anydipine-S(S-amlodipine) Tab. 2.5mg
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Telmisartan — Subjects assigned to the test group are oral administered Telmisartan 40 mg and S-Amlodopine 2.5 mg once a day for 12 weeks. However, if the blood pressure measured at 6 weeks after random allocation (Visit 3) is MSSBP ≥140 mmHg or MSDBP ≥ 90 mmHg, increase the dose to Telmisartan 80 mg for 6 weeks from Visit 3 to Visit 4 (End of study). However, if the need of dose increasing is not required according to the tester's judgment, the current dose can be maintained.
  Arms: Telmisartan
Drug: Losartan — Subjects assigned to the control group are oral administered Losartan 50 mg and S-Amlodopine 2.5 mg once a day for 12 weeks. However, if the blood pressure measured at 6 weeks after random allocation (Visit 3) is MSSBP ≥140 mmHg or MSDBP ≥ 90 mmHg, increase the dose to Losartan 100 mg for 6 weeks from Visit 3 to Visit 4 (End of study). However, if the need of dose increasing is not required according to the tester's judgment, the current dose can be maintained.
  Arms: Losartan

SUMMARY:
This is a multi-center, randomized, open-label, active comparator-controlled, phase 4 clinical trial to evaluate the blood pressure control of Telmisartan or Losartan in essential hypertensive patients with metabolic syndrome

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1 ratio to the following group; the test group [Telmisartan 40 mg + S-Amlodopine 2.5 mg], the control group [Losartan 50 mg + S-Amlodopine 2.5 mg]. If the blood pressure measured at 6 weeks time (Visit 3) based on the random allocation date (Visit 2) is MSSBP ≥140 mmHg or MSDBP ≥90 mmHg, the test group will increase the Telmisartan 80 mg, the control group will increase the dose to 100 mg for 6 weeks from Visit 3 to Visit 4(End of study). However, if the need of dose increasing is not required according to the investigator's judgment, the current dose can be maintained. All clinical trial drugs are administered orally once a day, and it is recommended to be administered at the same time(am) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

[Screening/Run-in period (Visit 1)]

* Adults over 19 years of age
* Patients who have been diagnosed with essential hypertension or who are taking antihypertensive drugs after diagnosis (However, if you are already taking antihypertensive drugs, you can discontinue/change the antihypertensive drugs and agree to this)
* At the time of screening/introduction (Visit 1), the following metabolic syndrome diagnosis criteria ①~④ satisfy ① fasting blood glucose standards, and those who meet at least one of ②~④ criteria (① Fasting blood sugar: ≥100 mg/dL or a state in which medication is being administered to control blood sugar, ② Waist circumference: male ≥90 cm, female ≥85 cm, ③ HDL-cholesterol: male <40 mg/dL, female <50 mg/dL or taking medication to increase HDL-cholesterol, ④ Triglyceride: ≥150 mg/dL or taking medication to lower triglyceride)

[Randomization (Visit 2)]

* Patients whose average sitting systolic or diastolic blood pressure measured in the arm selected as the reference arm during the screening test at the time of randomization (Visit 2) corresponds to the following

  * 140 mmHg ≤ mean sitting systolic blood pressure (MSSBP) < 180 mmHg
  * 90 mmHg ≤ mean sitting diastolic blood pressure (MSDBP) < 110 mmHg
* At the time of randomization (Visit 2), the following metabolic syndrome diagnosis criteria ① to ④ satisfy ① fasting blood sugar criteria, and those who meet at least one of ② to ④ criteria (① Fasting blood sugar: ≥100 mg/dL or a state in which medication is being administered to control blood sugar, ② Waist circumference: male ≥90 cm, female ≥85 cm, ③ HDL-cholesterol: male <40 mg/dL, female <50 mg/dL or taking medication to increase HDL-cholesterol, ④ Triglyceride: ≥150 mg/dL or taking medication to lower triglyceride)

Exclusion Criteria:

* Patients whose blood pressure measured at the time of screening/introduction (Visit 1) corresponds to any of the following

  * Patients with MSSBP ≥180 mmHg or MSDBP ≥110 mmHg
  * Patients with MSSBP ≥20 mmHg and MSDBP ≥10 mmHg difference in blood pressure measured 3 times in each arm
* Patients with a history of secondary hypertension or suspected secondary hypertension (aortic coarctation, hyperaldosteronemia, renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.)
* Patients with orthostatic hypotension with symptoms
* Patients with type 1 diabetes or poorly controlled diabetes (HbA1c >9.0%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
MSSBP change | Baseline (Visit 2), 12 weeks (Visit 4)
  MSSBP change between administration groups after 12 weeks (Visit 4) compared to baseline (Visit 2)

SECONDARY OUTCOMES:
MSSBP change | Baseline (Visit 2), 6 weeks (Visit 3)
  MSSBP change between administration groups after 6 weeks (Visit 3) compared to baseline (Visit 2)
MSDBP change | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  MSDBP change between administration groups compared to baseline (Visit 2) after 6 weeks (Visit 3) and 12 weeks (Visit 4)
Blood pressure normalization ratio | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Blood pressure normalization ratio (ratio of subjects with MSSBP <140 mmHg and MSDBP <90 mmHg) after 6 weeks (Visit 3) and 12 weeks (Visit 4) compared to baseline (Visit 2) between administration groups
Blood pressure response rate | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Blood pressure response rate (MSSBP reduction ≥20 mmHg and MSDBP reduction ≥10 mmHg) after 6 weeks (Visit 3) and 12 weeks (Visit 4) compared to baseline (Visit 2) between treatment groups
Changes in HOMA-IR | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Changes in HOMA-IR[(Fasting insulin(mU/L)×Fasting glucose(nmol/L))/22.5]
Changes in HOMA-β | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Changes in HOMA-β[(20×Fasting insulin(mU/L))/(Fasting glucose(nmol/L)-3.5)]
Changes in Glucose | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Changes in Glucose(nmol/L)
Changes in Insulin | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Changes in Insulin(mU/L) after 6 weeks (Visit 3) and 12 weeks (Visit 4) compared to baseline (Visit 2) between administration groups
Changes in HbA1c | Baseline (Visit 2), 6 weeks (Visit 3), 12 weeks (Visit 4)
  Changes in HbA1c (%) after 6 weeks (Visit 3) and 12 weeks (Visit 4) compared to baseline (Visit 2) between administration groups

CONTACTS AND LOCATIONS:
Overall Officials: Soo MD, MD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No